CLINICAL TRIAL: NCT06580860
Title: Psychiatric Multi-omics and Neuroimaging Project Database
Brief Title: Psychiatric Multi-omics and Neuroimaging Project
Acronym: PMNP
Status: Recruiting | Type: Observational
Sponsor: mingjun Zhong (Other)
Responsible Party: Sponsor-Investigator, mingjun Zhong, Principal Investigator, Second Xiangya Hospital of Central South University
Organization: Second Xiangya Hospital of Central South University (Other)
Other Study IDs: NSFC82201664
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Mental Disorders; Healthy Control
Keywords: schizophrenia; major depressive disorder; autism spectrum disorder; bipolar disorder; magnetic resonance imaging; multi-omics
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Depressive Disorder, Major; Autism Spectrum Disorder; Bipolar Disorder | interventions — Antipsychotic Agents; Antidepressive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10ml peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- PMNP-Healthy Norms: Healthy Norms
  Interventions: Drug: Antipsychotic drugs, antidepressants, mood stabilizers, and sleep aids
- PMNP-Subclinical high-risk: Subclinical high-risk
  Interventions: Drug: Antipsychotic drugs, antidepressants, mood stabilizers, and sleep aids
- PMNP-Schizophrenia and Psychosis: Schizophrenia and Psychosis patient
  Interventions: Drug: Antipsychotic drugs, antidepressants, mood stabilizers, and sleep aids
- PMNP-MDD: major depressive disorder patient
  Interventions: Drug: Antipsychotic drugs, antidepressants, mood stabilizers, and sleep aids
- PMNP-ASD: autism spectrum disorder patient
  Interventions: Drug: Antipsychotic drugs, antidepressants, mood stabilizers, and sleep aids
- PMNP-BD: bipolar disorder patient
  Interventions: Drug: Antipsychotic drugs, antidepressants, mood stabilizers, and sleep aids

INTERVENTIONS:
Drug: Antipsychotic drugs, antidepressants, mood stabilizers, and sleep aids — Patients with mental disorders should take the appropriate medicine as prescribed by the doctor，and the health norms are not required to take medicine.This study will not interfere with the medication regimen of doctors.

SUMMARY:
This study focuses on the structure and function of the brain and gene expression in peripheral blood of patients with schizophrenia, to explore the interaction and influence between the three. Patients with mental disorders who have been recruited will take their medication regularly for 1 year and participate in baseline and follow-up assessments.

DETAILED DESCRIPTION:
The study seeks to identify possible biological markers of schizophrenia and the effects of gene-environment interactions on brain structural and functional networks. So we can help doctors and scientific researchers better understand the neuropathological basis of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Age: 13-35 years old(Patients with healthy siblings can be extended to 14-35 years of age)
* Course of disease: <24 months
* Priority is given to patients who have never taken medicine or duration of drug use < 2 weeks
* No nuclear magnetic contraindications.

Exclusion Criteria:

* Family history of psychotic disorders, history of psychoactive substances abuse, alcohol dependence, or nicotine dependence
* Have a major physical disease or infectious disease
* History of coma and serious neurological disease 4.MRI contraindications.

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients from inpatient and outpatient the second Xiangya Hosptial of Central South University, Healthy controls from community, school and street recruitment
Sampling Method: Probability Sample
Enrollment: 1899 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
cortical morphology | 40 minutes
  Data were obtained using magnetic resonance scans
target gene charaacteristics | 1 day
  10ml peripheral blood was extracted for gene analysis
scale scores | 90 minutes.
  The score of each dimension and the total score were calculated according to the scale.The scale includes three dimensions: negative symptom, positive symptom and general psychopathology, and the score range of each dimension is different. The total score ranges from 30 to 210, with higher scores indicating worse results.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Xiangya hospital of central south univerity, Changsha, Hunan, China